CLINICAL TRIAL: NCT03496168
Title: An Open-Label Extension Study of Mavacamten (MYK-461) in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy Previously Enrolled in Study MYK-461-004 (PIONEER)
Brief Title: Extension Study of Mavacamten (MYK-461) in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy Previously Enrolled in PIONEER
Acronym: PIONEER-OLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV027-008
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Symptomatic; Obstructive; Left ventricular outflow tract gradient
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mavacamten (MYK-461) (Experimental)
  Interventions: Drug: mavacamten

INTERVENTIONS:
Drug: mavacamten — mavacamten capsules
  Other Names: MYK-461

SUMMARY:
This is a multicenter open-label study of the administration of mavacamten in participants with symptomatic obstructive HCM (oHCM) who previously participated in study MYK-461-004 (PIONEER-HCM).

ELIGIBILITY:
Key Inclusion Criteria:

* Completed Study MYK-461-004. Prior participation in a non-interventional observational study is allowed.
* Body weight > 45 kg at Screening
* Has safety laboratory parameters (chemistry and hematology) within normal limits

Key Exclusion Criteria:

* Has QTcF > > 500 ms or any other ECG abnormality considered by the investigator to pose a risk to subject safety (eg, second degree atrioventricular block type II)
* Since enrollment into Study MYK-461-004, has developed obstructive coronary artery disease (> 70% stenosis in one or more arteries) or known moderate or severe aortic valve stenosis
* Since enrollment into Study MYK-461-004, has developed any acute or serious comorbid condition (eg, major infection or hematologic, renal, metabolic, gastrointestinal, or endocrine dysfunction) that, in the opinion of the investigator or medical monitor, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Since enrollment into Study MYK-461-004 has developed clinically significant malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 0003, Scottsdale, Arizona
  - Local Institution - 0001, New Haven, Connecticut
  - Local Institution - 0004, Durham, North Carolina
  - Local Institution - 0002, Portland, Oregon

REFERENCES:
- [Derived] Masri A, Lester SJ, Stendahl JC, Hegde SM, Sehnert AJ, Balaratnam G, Shah A, Fox S, Wang A. Long-Term Safety and Efficacy of Mavacamten in Symptomatic Obstructive Hypertrophic Cardiomyopathy: Interim Results of the PIONEER-OLE Study. J Am Heart Assoc. 2024 Apr 16;13(8):e030607. doi: 10.1161/JAHA.123.030607. Epub 2024 Apr 9. PMID 38591260
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 Participants enrolled and treated
Groups:
- Mavacamtem: Mavacamtem
Period: Overall Study
Arm/Group | Mavacamtem
Started | 13
Completed | 11
Not Completed | 2
Not completed — Other Reasons | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Treatment Emergent Serious Adverse Events
Description: AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment.
  An SAE is defined as any untoward medical occurrence at any dose that:
  * Results in death
  * Is immediately life-threatening (places the participant at immediate risk of death from the event as it occurred)
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions
  * Results in a congenital abnormality or birth defect
  * Is an important medical event that may not result in death, be life- threatening, or require hospitalization, but may be considered an SAE when, based upon appropriate medical judgment, it may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: From first dose to end of treatment + 56 days (Approximately an average of 240 Weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  TEAEs | 13
  TESAEs | 5

2. Primary Outcome: Number of Participants Who Had Cardiovascular Death
Description: Number of participants who had died due to cardiovascular reasons.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

3. Primary Outcome: Number of Participants Who Experienced Sudden Death
Description: Number of participants who experienced sudden death
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

4. Primary Outcome: Number of Participants Who Were Hospitalized for Cardiovascular Reasons.
Description: Number of participants who were hospitalized for cardiovascular reasons.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 1

5. Primary Outcome: Number of Participants With Heart Failure Due to Systolic Dysfunction, Defined as Asymptomatic LVEF < 50%
Description: Number of participants with heart failure due to systolic dysfunction, defined as asymptomatic LVEF < 50%
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

6. Primary Outcome: Number of Participants With LVEF < 50% as Measured by Echocardiography.
Description: Number of participants with LVEF < 50% as measured by echocardiography.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 2

7. Primary Outcome: Number of Participants Who Were Experienced Myocardial Infarction
Description: Number of participants who experienced myocardial infarction.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

8. Primary Outcome: Number of Participants With Ventricular Arrhythmias.
Description: Types of Ventricular Arrhythmias measured in this endpoint will be:
  Ventricular Tachycardia Ventricular Fibrilation Ventricular Flutter
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Ventricular Tachycardia | 1
  Ventricular Fibrilation | 0
  Ventricular Flutter | 0
  Torsades De Pointe | 0

9. Primary Outcome: Number of Participants Who Experienced Syncope
Description: Number of participants who experienced syncope.
  Syncope will be defined as participants who experienced dizziness or orthostatic hypotension.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Dizziness | 2
  Orthostatic Hypotension | 1

10. Primary Outcome: Number of Participants Who Experienced Seizures
Description: Number of participants who were experienced seizures.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

11. Primary Outcome: Number of Participants Who Were Experienced Strokes
Description: Number of participants who were experienced strokes.
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

12. Primary Outcome: Number of Participants With a Change in QT and QTcF Intervals.
Description: Number of participants with a change in QTcF intervals.
  QTcF: An electrocardiographic finding in which the QT interval corrected for heart rate using Fridericia's formula. QTc = QT/∛(RR/1000)
  RR = Respiration rate
  QT Interval: Ventricular depolarization plus ventricular repolarization Normal Range: 400 to 460 msec
Time Frame: From first dose to end of study, (approximately 260 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Post Baseline QTcF > 450msec | 7
  Post Baseline QTcF > 480msec | 1
  Post Baseline QTcF > 500msec | 1
  Change from Baseline QTcF > 30 msec | 2
  Change from Baseline QTcF > 60 msec | 1

13. Primary Outcome: Post-exercise Left Ventricular Outflow Tract (LVOT) Gradient Over Time
Description: Number of participants with changes of Post-exercise left ventricular outflow tract (LVOT) gradient over time
Time Frame: At Baseline, Week 4, Week 48, Week 72, Week 156, Week 204 and Week 252
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Baseline: < 30 mmHg | 0
  Baseline: >= 30 mmHg to < 50 mmHg | 0
  Baseline: >= 50 mmHg | 13
  Week 4: < 30 mmHg | 0
  Week 4: >= 30 mmHg to < 50 mmHg | 3
  Week 4: >= 50 mmHg | 10
  Week 48: number analyzed (Participants) | 11
  Week 48: < 30 mmHg | 6
  Week 48: >= 30 mmHg to < 50 mmHg | 3
  Week 48: >= 50 mmHg | 2
  Week 72: number analyzed (Participants) | 11
  Week 72: < 30 mmHg | 8
  Week 72: >= 30 mmHg to < 50 mmHg | 0
  Week 72: >= 50 mmHg | 3
  Week 156: number analyzed (Participants) | 12
  Week 156: < 30 mmHg | 10
  Week 156: >= 30 mmHg to < 50 mmHg | 0
  Week 156: >= 50 mmHg | 2
  Week 204: number analyzed (Participants) | 12
  Week 204: < 30 mmHg | 9
  Week 204: >= 30 mmHg to < 50 mmHg | 1
  Week 204: >= 50 mmHg | 2
  Week 252: number analyzed (Participants) | 11
  Week 252: < 30 mmHg | 9
  Week 252: >= 30 mmHg to < 50 mmHg | 0
  Week 252: >= 50 mmHg | 2

14. Primary Outcome: Resting Left Ventricular Outflow Tract (LVOT) Gradient Over Time
Description: Resting left ventricular outflow tract (LVOT) gradient over time
Time Frame: At Baseline, Week 4, Week 48, Week 72, Week 156, Week 204 and Week 252
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Baseline: < 30 mmHg | 3
  Baseline: >= 30 mmHg to < 50 mmHg | 2
  Baseline: >= 50 mmHg | 8
  Week 4: < 30 mmHg | 8
  Week 4: >= 30 mmHg to < 50 mmHg | 0
  Week 4: >= 50 mmHg | 5
  Week 48: number analyzed (Participants) | 12
  Week 48: < 30 mmHg | 11
  Week 48: >= 30 mmHg to < 50 mmHg | 1
  Week 48: >= 50 mmHg | 0
  Week 72: number analyzed (Participants) | 11
  Week 72: < 30 mmHg | 11
  Week 72: >= 30 mmHg to < 50 mmHg | 0
  Week 72: >= 50 mmHg | 0
  Week 156: number analyzed (Participants) | 12
  Week 156: < 30 mmHg | 11
  Week 156: >= 30 mmHg to < 50 mmHg | 1
  Week 156: >= 50 mmHg | 0
  Week 204: number analyzed (Participants) | 12
  Week 204: < 30 mmHg | 10
  Week 204: >= 30 mmHg to < 50 mmHg | 1
  Week 204: >= 50 mmHg | 1
  Week 252: number analyzed (Participants) | 11
  Week 252: < 30 mmHg | 11
  Week 252: >= 30 mmHg to < 50 mmHg | 0
  Week 252: >= 50 mmHg | 0

15. Primary Outcome: Post Valsalva Left Ventricular Outflow Tract (LVOT) Gradient Over Time
Description: Post Valsalva left ventricular outflow tract (LVOT) gradient over time
Time Frame: At Baseline, Week 4, Week 48, Week 72, Week 156, Week 204 and Week 252
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants
  Baseline: number analyzed (Participants) | 12
  Baseline: < 30 mmHg | 0
  Baseline: >= 30 mmHg to < 50 mmHg | 1
  Baseline: >= 50 mmHg | 11
  Week 4: < 30 mmHg | 3
  Week 4: >= 30 mmHg to < 50 mmHg | 2
  Week 4: >= 50 mmHg | 8
  Week 48: number analyzed (Participants) | 12
  Week 48: < 30 mmHg | 9
  Week 48: >= 30 mmHg to < 50 mmHg | 1
  Week 48: >= 50 mmHg | 2
  Week 72: number analyzed (Participants) | 11
  Week 72: < 30 mmHg | 9
  Week 72: >= 30 mmHg to < 50 mmHg | 1
  Week 72: >= 50 mmHg | 1
  Week 156: number analyzed (Participants) | 12
  Week 156: < 30 mmHg | 10
  Week 156: >= 30 mmHg to < 50 mmHg | 1
  Week 156: >= 50 mmHg | 1
  Week 204: number analyzed (Participants) | 12
  Week 204: < 30 mmHg | 9
  Week 204: >= 30 mmHg to < 50 mmHg | 0
  Week 204: >= 50 mmHg | 3
  Week 252: number analyzed (Participants) | 11
  Week 252: < 30 mmHg | 10
  Week 252: >= 30 mmHg to < 50 mmHg | 0
  Week 252: >= 50 mmHg | 1

16. Primary Outcome: Participants With >= 1 NYHA Function Class Improvement
Description: Participants with >= 1 NYHA function class improvement.
  The NYHA Functional Classification of heart failure assigns participants to 1 of 4 categories based on the participant's symptoms.
  Class 1: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  Class 2: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class 3: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class 4: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: At Baseline, Week 4, Week 8, Week 24, Week 48, Week 72, Week 96, Week 120, Week 144, Week 156, Week 180, Week 204, Week 228 and Week 252
Population: Safety Analysis Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Percentage of Participants
  Change from baseline at week 4 | 15.4 [1.92 to 45.45]
  Change from baseline at week 8 | 46.2 [19.22 to 74.87]
  Change from baseline at week 24 | 76.9 [46.19 to 94.96]
  Change from baseline at week 48: number analyzed (Participants) | 12
  Change from baseline at week 48 | 75.0 [42.81 to 94.51]
  Change from baseline at week 72: number analyzed (Participants) | 11
  Change from baseline at week 72 | 90.9 [58.72 to 99.77]
  Change from baseline at week 96: number analyzed (Participants) | 12
  Change from baseline at week 96 | 83.3 [51.59 to 97.91]
  Change from baseline at week 120: number analyzed (Participants) | 12
  Change from baseline at week 120 | 91.7 [61.52 to 99.79]
  Change from baseline at week 144: number analyzed (Participants) | 12
  Change from baseline at week 144 | 91.7 [61.52 to 99.79]
  Change from baseline at week 156: number analyzed (Participants) | 12
  Change from baseline at week 156 | 91.7 [61.52 to 99.79]
  Change from baseline at week 180: number analyzed (Participants) | 12
  Change from baseline at week 180 | 83.3 [51.59 to 97.91]
  Change from baseline at week 204: number analyzed (Participants) | 12
  Change from baseline at week 204 | 83.3 [51.59 to 97.91]
  Change from baseline at week 228: number analyzed (Participants) | 12
  Change from baseline at week 228 | 83.3 [51.59 to 97.91]
  Change from baseline at week 252: number analyzed (Participants) | 11
  Change from baseline at week 252 | 90.9 [58.72 to 99.77]

17. Primary Outcome: Mean Change From Baseline in the Overall KCCQ PRO Score.
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self-administered 23-item questionnaire questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. Overall KCCQ Pro score is the average of all the domains, symptom frequency and symptom burden scores, and transformed to a single score which ranged from 0 (worst) to 100 (the best possible status), where the higher score reflected better health status.
Time Frame: as for outcome 16
Population: Safety Analysis Population
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Scores on a Scale
  Change from baseline at week 4 | 5.809 (8.7200)
  Change from baseline at week 8 | 12.304 (15.7392)
  Change from baseline at week 24 | 16.931 (18.4502)
  Change from baseline at week 48: number analyzed (Participants) | 12
  Change from baseline at week 48 | 16.345 (18.2986)
  Change from baseline at week 72: number analyzed (Participants) | 11
  Change from baseline at week 72 | 18.600 (16.7875)
  Change from baseline at week 96: number analyzed (Participants) | 12
  Change from baseline at week 96 | 16.162 (18.2376)
  Change from baseline at week 120: number analyzed (Participants) | 12
  Change from baseline at week 120 | 18.142 (15.9249)
  Change from baseline at week 144: number analyzed (Participants) | 12
  Change from baseline at week 144 | 17.860 (15.5829)
  Change from baseline at week 156: number analyzed (Participants) | 12
  Change from baseline at week 156 | 18.750 (15.5701)
  Change from baseline at week 180: number analyzed (Participants) | 12
  Change from baseline at week 180 | 16.674 (15.6328)
  Change from baseline at week 204: number analyzed (Participants) | 12
  Change from baseline at week 204 | 19.661 (15.9783)
  Change from baseline at week 228: number analyzed (Participants) | 11
  Change from baseline at week 228 | 91.122 (10.6882)
  Change from baseline at week 252: number analyzed (Participants) | 11
  Change from baseline at week 252 | 89.489 (12.7977)

18. Primary Outcome: Mean Change From Baseline in Serum NT-proBNP.
Description: Mean change from baseline in Serum N-terminal pro B-type natriuretic peptide levels.
Time Frame: as for outcome 16
Population: Safety Analysis Population
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
ng/L
  Change from baseline at week 4 | -1017.4 (1540.78)
  Change from baseline at week 8 | -1440.6 (2063.89)
  Change from baseline at week 24 | -1512.8 (2242.40)
  Change from baseline at week 48: number analyzed (Participants) | 12
  Change from baseline at week 48 | -1579.2 (2328.81)
  Change from baseline at week 72: number analyzed (Participants) | 11
  Change from baseline at week 72 | -1708.4 (2448.93)
  Change from baseline at week 96: number analyzed (Participants) | 12
  Change from baseline at week 96 | -1579.1 (2339.95)
  Change from baseline at week 120: number analyzed (Participants) | 11
  Change from baseline at week 120 | -1692.7 (2426.02)
  Change from baseline at week 144: number analyzed (Participants) | 12
  Change from baseline at week 144 | -1507.8 (2407.34)
  Change from baseline at week 156: number analyzed (Participants) | 11
  Change from baseline at week 156 | -1673.5 (2460.82)
  Change from baseline at week 180: number analyzed (Participants) | 12
  Change from baseline at week 180 | -1433.6 (2347.72)
  Change from baseline at week 204: number analyzed (Participants) | 12
  Change from baseline at week 204 | -1568.7 (2400.63)
  Change from baseline at week 228: number analyzed (Participants) | 11
  Change from baseline at week 228 | -1325.5 (2368.77)
  Change from baseline at week 252: number analyzed (Participants) | 11
  Change from baseline at week 252 | -1681.5 (2409.67)

19. Primary Outcome: Number of Participants Who Received Septal Reduction Therapy
Description: Number of participants who received septal reduction therapy
Time Frame: 252 weeks
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
Participants | 0

20. Primary Outcome: Plasma Concentration of Mavacamen Overtime
Description: Plasma concentration of Mavacamen overtime
Time Frame: as for outcome 16
Population: PK Analysis Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mavacamtem
Number analyzed (Participants) | 13
ng/mL
  Week 4 | 166.51 (32.1)
  Week 8 | 334.65 (21.5)
  Week 24 | 396.18 (31.7)
  Week 48: number analyzed (Participants) | 12
  Week 48 | 400.15 (35.1)
  Week 72: number analyzed (Participants) | 11
  Week 72 | 407.27 (24.4)
  Week 96: number analyzed (Participants) | 12
  Week 96 | 422.82 (29.3)
  Week 120: number analyzed (Participants) | 11
  Week 120 | 399.17 (33.2)
  Week 144: number analyzed (Participants) | 10
  Week 144 | 410.23 (42.8)
  Week 156: number analyzed (Participants) | 12
  Week 156 | 400.02 (44.1)
  Week 180: number analyzed (Participants) | 12
  Week 180 | 265.04 (57.9)
  Week 204: number analyzed (Participants) | 12
  Week 204 | 376.25 (69.5)
  Week 228: number analyzed (Participants) | 11
  Week 228 | 355.29 (72.3)
  Week 252: number analyzed (Participants) | 12
  Week 252 | 334.57 (52.1)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 56 days): Approximately 240 Weeks All-Cause mortality (From randomization to end of study): Approximately 260 Weeks
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Mavacamten: Mavacamtem
Arm/Group | Mavacamten
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=13)
Mitral valve incompetence (Cardiac disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Aortic stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mavacamten (N=13)
Leukocytosis (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac flutter (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 5
Oedema peripheral (General disorders) | 1
Peripheral swelling (General disorders) | 1
Biliary obstruction (Hepatobiliary disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 1
Prostate infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Cortisol decreased (Investigations) | 1
Drug level increased (Investigations) | 2
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 1
Troponin increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Insulin resistance (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cluster headache (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dizziness exertional (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 3
Facial spasm (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Ophthalmic migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Essential hypertension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03496168/Prot_SAP_000.pdf